CLINICAL TRIAL: NCT02906618
Title: An Absolute Bioavailability Study of LY3039478 in Healthy Subjects Using the Intravenous Tracer Method
Brief Title: Study of LY3039478 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16344; I6F-MC-JJCG (Other: Eli Lilly and Company); 2016-001073-33 (EudraCT Number)
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Results first posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Healthy
MeSH Terms: interventions — crenigacestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY3039478 - Oral (Experimental): LY3039478 given once, orally
  Interventions: Drug: LY3039478
- 13C 15N 2H-LY3039478 - IV (Experimental): 13C 15N 2H-LY3039478 given once, IV
  Interventions: Drug: 13C 15N 2H-LY3039478 IV

INTERVENTIONS:
Drug: LY3039478 — Administered orally
  Arms: LY3039478 - Oral
Drug: 13C 15N 2H-LY3039478 IV — Administered IV
  Arms: 13C 15N 2H-LY3039478 - IV

SUMMARY:
The study involves one dose of LY3039478 given by mouth followed by an intravenous infusion (IV) (via a tube linked to a small needle in the vein) of LY3039478. The results of this study will help to answer the following research questions:

* How much LY3039478 gets into the blood stream when given by mouth as a capsule compared to when given by an IV
* How long it takes the body to remove the study drug
* The safety of LY3039478 and any side effects that might be associated with it

Participation in the study is expected to last up to 7 weeks. There will be screening, a single study period, and a follow-up.

ELIGIBILITY:
Inclusion Criteria:

- Have a body mass index (BMI) of 18.5 to 32.0 kilogram per meter square (kg/m²) inclusive

Exclusion Criteria:

- Have previously completed or withdrawn from this study or any other study investigating LY3039478, and have previously received the investigational product

• Have known allergies to LY3039478, related compounds or any components of the formulation, or history of significant atopy in the opinion of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-10-04; Primary Completion 2016-11-11 (Actual); Study Completion 2016-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Leeds, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- LY3039478 - Oral and 13C 15N 2H-LY3039478 - IV: Simultaneous administration of a single oral dose of 75 milligram (mg) of LY3039478 and a 45-minute IV administration of 350 microgram (μg) 13C15N2H-LY3039478 in healthy participants.
Period: Overall Study
Arm/Group | LY3039478 - Oral and 13C 15N 2H-LY3039478 - IV
Started | 12
Received at Least One Dose of Study Drug | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: LY3039478 given once, orally and 13C 15N 2H-LY3039478 given once, IV.
Arm/Group | Overall
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 12
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 177.00 (7.41)
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 80.97 (10.00)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram/square meter (kg/m²)] | 25.82 (2.50)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) From Time Zero to the Last Time Point With a Measurable Concentration (AUC[0-tlast]) of LY3039478 and 13C 15N 2H-LY3039478
Description: Pharmacokinetics (PK) is the area under the concentration versus time curve (AUC) from time zero to the last time point with a measurable concentration (AUC[0-tlast]) of LY3039478 and 13C 15N 2H-LY3039478.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3.5, 4, 6, 8, 12, 24, 36, 48 Hours Postdose
Population: All participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nangogram*hour/milliliter (ng*h/mL)
Groups:
- LY3039478 - Oral: On Day 1 following an overnight fast of at least 10 hours, participants received a single oral dose of 75 mg LY3039478.
- 13C 15N 2H-LY3039478 - IV: On Day 1, 15 minutes after the 75 mg oral dose of unlabeled LY3039478, an IV infusion (duration 45 minutes) of 350 μg 13C 15N 2H-LY3039478 was started.
Arm/Group | LY3039478 - Oral | 13C 15N 2H-LY3039478 - IV
Number analyzed (Participants) | 12 | 12
nangogram*hour/milliliter (ng*h/mL) | 1920 (23) | 15.6 (16)

2. Primary Outcome: PK: AUC From Zero to Infinity (AUC[0 - Inf]) of LY3039478 and 13C 15N 2H-LY3039478
Description: PK is AUC from zero to infinity (AUC[0 - inf]) of LY3039478 and 13C 15N 2H-LY3039478.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3.5, 4, 6, 8, 12, 24, 36, 48 Hours Postdose
Population: All participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | LY3039478 - Oral | 13C 15N 2H-LY3039478 - IV
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 1920 (23) | 15.6 (16)
Statistical Analysis 1: Comparison: LY3039478 - Oral vs 13C 15N 2H-LY3039478 - IV; Test type: Other — A mixed-effect analysis of variance model was applied to the log-transformed dose-adjusted AUC(0-∞) of LY3039478 after oral dosing and IV administration of 13C 15N 2H-LY3039478. The model contained a fixed effect for formulation (oral or IV) and a random effect for participant; Ratio of geometric LS means = 0.572, 90% CI 2-sided [0.532 to 0.615]

3. Secondary Outcome: PK: Maximum Observed Drug Concentration (Cmax) of LY3039478 and 13C 15N 2H-LY3039478 - IV
Description: PK is the maximum observed drug concentration (cmax) of LY3039478 13C 15N 2H-LY3039478 - IV.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3.5, 4, 6, 8, 12, 24, 36, 48 Hours Postdose
Population: All participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/millilter (ng/mL)
Arm/Group | LY3039478 - Oral | 13C 15N 2H-LY3039478 - IV
Number analyzed (Participants) | 12 | 12
nanogram/millilter (ng/mL) | 444 (23) | 7.24 (15)

4. Secondary Outcome: PK: Time of Cmax (Tmax) of LY3039478 and 13C 15N 2H-LY3039478
Description: PK is the time of Cmax (tmax) of LY3039478 and 13C 15N 2H-LY3039478.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3.5, 4, 6, 8, 12, 24, 36, 48 Hours Postdose
Population: All participants who received at least one dose of study drug.
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | LY3039478 - Oral | 13C 15N 2H-LY3039478 - IV
Number analyzed (Participants) | 12 | 12
hour (hr) | 1.500 [1.000 to 3.500] | 0.750 [0.750 to 0.750]

5. Secondary Outcome: PK: Half Life Associated With The Terminal Rate Constant (t1/2) of LY3039478 and 13C 15N 2H-LY3039478
Description: PK is the half life associated with the terminal rate constant (t1/2) of LY3039478 and 13C 15N 2H-LY3039478.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3.5, 4, 6, 8, 12, 24, 36, 48 Hours Postdose
Population: All participants who received at least one dose of study drug.
Measure: Geometric Mean (Full Range); unit: hr
Arm/Group | LY3039478 - Oral | 13C 15N 2H-LY3039478 - IV
Number analyzed (Participants) | 12 | 12
hr | 5.42 [4.93 to 6.88] | 3.31 [2.84 to 3.75]

ADVERSE EVENTS:
Groups:
- LY3039478 - Oral and 13C 15N 2H-LY3039478 - IV: Simultaneous administration of a single oral dose of 75 mg of LY3039478 and a 45-minute IV administration of 350 μg 13C 15N 2H-LY3039478 in healthy participants.
Arm/Group | LY3039478 - Oral and 13C 15N 2H-LY3039478 - IV
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3039478 - Oral and 13C 15N 2H-LY3039478 - IV (N=12)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days